CLINICAL TRIAL: NCT07403643
Title: Safety, Pharmacokinetics, and Preliminary Efficacy of Tafenoquine for the Treatment of Vivax Malaria in Papua New Guinean Children
Brief Title: Investigating the Pharmacology of Tafenoquine in Papua New Guinean Children With Uncomplicated Malaria
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES67418-B
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Uncomplicated Malaria
Keywords: tafenoquine; vivax malaria; radical cure; pharmacokinetics; children
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Tafenoquine + Artemether-Lumefantrine (Experimental): Single-dose tafenoquine as 10 mg/kg given with the first dose of artemether-lumefantrine treatment regimen (ARM 1.7 mg/kg and LUM 10 mg/kg, twice daily for 3 days) with water and a low-fat meal
  Interventions: Drug: Single dose tafenoquine (10 mg/kg); Drug: Artemether + Lumefantrine
- Group B: Tafenoquine + Dihydroartemisinin-piperaquine (Experimental): Single-dose tafenoquine as 10 mg/kg given with the first dose of dihydroartemisinin-piperaquine (DHA 2.5 mg/kg and PQ phosphate 20 mg/kg, once daily for 3 days) with water and a low-fat meal
  Interventions: Drug: Single dose tafenoquine (10 mg/kg); Drug: Dihydroartemisinin-piperaquine (DHA-PPQ)

INTERVENTIONS:
Drug: Single dose tafenoquine (10 mg/kg) — Participants will receive single-dose TQ as 10 mg/kg given with the first dose of ACT. Food (low-fat meal) is taken to attenuate any gastrointestinal adverse effects that are related to taking TQ on an empty stomach. Combinations of full or half-tablets will be swallowed whole or crushed lightly (tablets) or dissolved in boiled water (if dispersible tablets are available), as directly observed treatment. Children vomiting within the first 30 minutes of treatment will be withdrawn, and will receive the remaining treatment course of their randomized ACT as for PNG Standard Treatment Guidelines.
  Other Names: Tafenoquine succinate; TQ; Kodatef
Drug: Dihydroartemisinin-piperaquine (DHA-PPQ) — Participants will receive dihydroartemisinin-piperaquine (DHA 2.5 mg/kg and PQ phosphate 20 mg/kg), once daily for 3 days with water and a low-fat meal. Combinations of full or half-tablets will be swallowed whole or crushed lightly (tablets) or dissolved in boiled water (if dispersible tablets are available), as directly observed treatment.
  Other Names: DP; DHA-PPQ; Eurartesim
  Arms: Group B: Tafenoquine + Dihydroartemisinin-piperaquine
Drug: Artemether + Lumefantrine — Participants will receive artemether-lumefantrine (ARM 1.7 mg/kg and LUM 10 mg/kg) twice daily for 3 days with water and a low-fat meal. Combinations of full or half-tablets will be swallowed whole or crushed lightly (tablets) or dissolved in boiled water (if dispersible tablets are available). Morning doses will be observed as directly observed treatment, with evening doses dispensed to the parent/guardian each day. Parents will be asked to report approximate time of evening dosing the following morning, and return any pills that were not successfully administered.
  Other Names: ARM-LUM; Mala1; Coartem
  Arms: Group A: Tafenoquine + Artemether-Lumefantrine

SUMMARY:
Plasmodium vivax is the most geographically widespread malaria species and the second largest contributor to symptomatic malaria worldwide. It accounts for half of all malaria cases outside Africa, with an estimated 14.3 million clinical vivax malaria cases reported annually, contributing to an annual cost of US$359 million. Children are most vulnerable to infection, with P. vivax prevalence peaking between 2 to 6 years of age. In Papua New Guinea (PNG), there are >1.5 million suspected P. vivax cases annually, and while P. falciparum infections are the most prevalent, P. vivax transmission is the most intense in the world. P. vivax in PNG provides a unique epidemiological setting in which to assess innovative treatments in children.The complex biology of P. vivax represents a challenge for malaria control and chemotherapy, especially dormant liver-stage parasites (hypnozoites) which can reactivate (relapse) and cause disease at a time remote from the primary infection. Hypnozoite relapse is the primary cause of vivax malaria in endemic regions and is resistant to most antimalarial drugs. Identifying effective treatments for radical cure, the complete elimination of parasites (both blood- and liver-stage), is therefore a priority. The World Health Organization (WHO) recommends a 14-day radical cure regimen for uncomplicated vivax malaria; comprised of blood stage treatment (chloroquine or artemisinin combination therapy (ACT)) and 14 days of the 8-aminoquinoline drug primaquine (PQ; 0.25-0.5 mg/kg/day) for liver-stage cure. More recently, the 8-aminoquinoline tafenoquine has garnered interest as an alternative radical cure agent to primaquine. However, there is limited data on the pharmacokinetics, tolerability and radical cure efficacy of tafenoquine in children. Furthermore, early data suggest a drug interaction between TQ and artemisinin combination therapy (ACT) drugs - which requires further investigation and confirmation. This study will generate critical paediatric safety, tolerability, pharmacokinetic, and preliminary efficacy data for TQ when administered with either artemether-lumefantrine or dihydroartemisinin-piperaquine in PNG children with uncomplicated malaria.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the safety, tolerability, pharmacokinetic disposition and preliminary efficacy of tafenoquine, when co-administered as part of a radical cure regimen with two artemisinin combination therapies in Papua New Guinean children with uncomplicated malaria. This study represents the second part of a multi-phase investigation of tafenoquine in PNG children (Study 1: NCT07052162). In this study, children aged 2 to 12 years will be eligible for inclusion in the study providing they have uncomplicated malaria (P. falciparum and/or P. vivax malaria; confirmed by rapid diagnostic test and/or microscopy), normal G6PD activity (>70% enzyme activity by SD Biosensor), no evidence of severe malaria, no significant comorbidity, and no history of previous hypersensitivity to 8-aminoquinolines, artemether-lumefantrine or dihydroartemisinin-piperaquine. All participants will be admitted to the Alexishafen Health Centre for the first 24-hours of the study, to facilitate blood sampling and clinical monitoring. After admission, baseline demographic and medical history will be taken, and the participants will undergo a full clinical assessment to establish baseline safety indices. The 60 participants will then be randomized 1:1 to receive either i) single-dose TQ as 10 mg/kg given with the first dose of artemether-lumefantrine treatment regimen (Coartem®; ARM 1.7 mg/kg and LUM 10 mg/kg, twice daily for 3 days) with water and a low-fat meal (unless indicated otherwise in Study 1), or ii) single-dose TQ as 10 mg/kg given with the first dose of dihydroartemisinin-piperaquine (Eurartesim®; DHA 2.5 mg/kg and PQ phosphate 20 mg/kg, once daily for 3 days) with water and a low-fat meal (unless indicated otherwise in Study 1). For pharmacokinetic analysis, each participant will be allocated a randomised sampling schedule with dried blood spots for pharmacokinetic analysis performed at 6 of 15 time points (2, 4, 8, 12, 18, 24, 38 and 48 hours, Days 3, 4, 7, 14, 28, 42 and 56). At each allocated time point, 0.5 mL samples will be collected by finger-prick with five 50 µL blood drops spotted on to Whatman Protein 903 cards for dried blood spot analysis. The remaining blood will be collected into lithium heparin anticoagulant. Both dried blood spot and plasma samples will be collected at all time points for pharmacokinetic analyses. Standardised review, including adverse-effect questionnaires, and clinical monitoring (haemoglobin, methaemoglobin, reticulocyte counts, malaria blood films) will be conducted at all daily follow-up time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, 56 and 84). Safety testing (hepatorenal function tests (ALT, total bilirubin, creatinine), haemoglobin, urine dipstick analysis and electrocardiogram trace, will be taken at 4, 24 hours and on Days 3, 7 and 28.

The primary aim of the study is to characterise the pharmacokinetic profile of TQ (and its primary metabolite) in PNG children.

Secondary objectives include;

1. To assess the safety of TQ in PNG children
2. To assess the preliminary relapse efficacy of TQ given with artemether-lumefantrine.
3. To assess the preliminary relapse efficacy of TQ given with dihydroartemisinin-piperaquine.
4. To assess the tolerability of TQ in PNG children.

The investigators hypothesise that:

1. A single TQ 10 mg/kg dose is safe and efficacious for use in children with uncomplicated malaria.
2. TQ has no clinically relevant effects on the pharmacokinetics of artemether, lumefantrine, or their metabolites.
3. Cut or crushed tablets will not be well tolerated, although tolerability will improve with administration of whole tablets or dispersible tablets.

ELIGIBILITY:
Inclusion Criteria:

* Have normal G6PD activity (>70% enzyme activity) as confirmed by quantitative SD Biosensor
* Do not have severe malaria (by WHO criteria)
* Have rapid diagnostic test and/or microscopically confirmed uncomplicated malaria (any species)
* Have no significant co-morbidity
* Have no history of hypersensitivity to primaquine
* Have no history of hypersensitivity to artemether-lumefantrine or dihydroartemisinin-piperaquine
* Are able to attend all scheduled follow-up visits

Exclusion Criteria:

* Have <70% G6PD enzyme activity, as confirmed by quantitative SD Biosensor
* Have signs or symptoms of severe malaria (by WHO criteria)
* Test negative for malaria by rapid diagnostic test and/or microscopy
* Have signs or symptoms of a significant co-morbidity
* Have a history of hypersensitivity to primaquine
* Have a history of hypersensitivity to artemether-lumefantrine or dihydroartemisinin-piperaquine
* Cannot, or are not willing, to attend all scheduled follow-up visits

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: Tafenoquine terminal elimination half-life | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetic: Tafenoquine distribution half-life | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetic: Tafenoquine absorption half-life | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetics: Tafenoquine clearance | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetics: Tafenoquine volume of distribution | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetic: Tafenoquine maximal concentration | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.
Pharmacokinetics: Tafenoquine area under concentration-time curve | 56-days after tafenoquine administration
  Pharmacokinetic parameters of tafenoquine and 5,6-orthoquinone tafenoquine, will be ascertained using a nonlinear mixed-effects modelling approach (NONMEM), based on drug concentrations determined from blood samples collected at baseline (Day 0) and 6 of 13 randomized collection time points (2, 4, 8, 12, 24 and 48 hours and Days 3, 4, 7, 14, 28, 42 and 56.

SECONDARY OUTCOMES:
Safety: Change in haemoglobin over 84 days | 84-days from tafenoquine administration
  A fingerprick blood sample will be drawn at baseline to determine pre-treatment haemoglobin concentration (point-of-care HemoCue Hb201+, Radiometer, Australia). To monitor for post-treatment haemolysis, fingerprick haemoglobin samples will be taken at safety time points (4 and 24 hours, and on days 3, 7 and 28 post tafenoquine dosing) and all standardised review time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, 56 and 84).
Safety: Change in methaemoglobin over 28 days | 28-days from drug administration.
  Methaemoglobin will be assessed by a Rad57 pulse oximeter with SpMet function (Masimo, USA) at all defined safety time points (4 and 24 hours) and standardised review time points (Days 0, 1, 2, 3, 4, 7, 14, and 28).
Safety: Change in hepatorenal function over 28 days | 28-days from tafenoquine administration
  Hepatorenal function (creatinine, total bilirubin and alanine transaminase [ALT]) will be analysed on a Fuji Dri-Chem NX500 analyser (Fujifilm, Japan). 100 µL fingerprick blood samples will be collected at baseline, 4 and 24 hours, and on Days 3, 7 and 28 after tafenoquine dosing.
Safety: Change in rate corrected QTc over 28 days | 28-days from tafenoquine administration
  A 12-lead electrocardiogram will be conducted at baseline, 4 and 24 hours, and on Days 3, 7 and 28 after tafenoquine dosing to determine change in rate corrected QTc.
Efficacy: PCR adjusted Day-28 P. vivax relapse efficacy | 28-days from tafenoquine administration
  Blood smears for malarial microscopy and dried blood spots for molecular parasitology will be carried out at all daily follow-up time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, 56 and 84). All blood films for malarial microscopy will be examined by two skilled microscopists blinded to treatment. Slides discrepant for positivity/negativity, speciation or parasitaemia (>3x difference) will be adjudicated by a senior microscopist. Quantitative multi-species PCR will be assayed (using validated methods) on all collected samples to confirm outcomes from malarial microscopy, and report PCR adjusted relapse efficacy.
Efficacy: PCR adjusted Day-42 P. vivax relapse efficacy | 42-days from tafenoquine administration
  Blood smears for malarial microscopy and dried blood spots for molecular parasitology will be carried out at all daily follow-up time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, 56 and 84). All blood films for malarial microscopy will be examined by two skilled microscopists blinded to treatment. Slides discrepant for positivity/negativity, speciation or parasitaemia (>3x difference) will be adjudicated by a senior microscopist. Quantitative multi-species PCR will be assayed (using validated methods) on all collected samples to confirm outcomes from malarial microscopy, and report PCR adjusted relapse efficacy.
Efficacy: PCR adjusted Day-84 P. vivax relapse efficacy | 84-days after tafenoquine administration
  Blood smears for malarial microscopy and dried blood spots for molecular parasitology will be carried out at all daily follow-up time points (Days 0, 1, 2, 3, 4, 7, 14, 28, 42, 56 and 84). All blood films for malarial microscopy will be examined by two skilled microscopists blinded to treatment. Slides discrepant for positivity/negativity, speciation or parasitaemia (>3x difference) will be adjudicated by a senior microscopist. Quantitative multi-species PCR will be assayed (using validated methods) on all collected samples to confirm outcomes from malarial microscopy, and report PCR adjusted relapse efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Brioni R Moore, PhD, Principal Investigator — Curtin University
Locations (1):
- Alexishafen Health Centre, Madang, Madang Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: No
Data may be shared upon contact with the principal investigators and approval by the PNG Institute of Medical Research. This process will be conducted on a case by case basis, as per agreements between collaborative partners.